CLINICAL TRIAL: NCT01561820
Title: Community-based, Buddy-supported Exercise in Patients With MCI: a Pilot Trial
Brief Title: Mild Cognitive Impairment, Buddy Supported Exercise/ My Buddy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00018495
Record Dates: First submitted 2012-03-08; First posted 2012-03-23 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment; Cognitive Disorders
Keywords: mild cognitive impairment; cognitive disorders; exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buddy (Active Comparator): Participant will be assigned a buddy that will meet with them at the gym for each of their exercise sessions. This person will serve as a source of support and motivation for them and will also help them remember and stick to the goals set for you. This person will also help them maintain their exercise logs and ensure they are correct. The buddy will not be exercising with them, but will just be there with them while you exercise.
  Interventions: Behavioral: 5-month aerobic exercise intervention
- Non Buddy (Placebo Comparator): Participants will not be assigned a buddy (and are not allowed to bring someone with them as a buddy). They will be asked to exercise on their own and remember the goals set for them. They will also be responsible for filling out their own exercise logs and ensuring they are correct.
  Interventions: Behavioral: 5-month aerobic exercise intervention

INTERVENTIONS:
Behavioral: 5-month aerobic exercise intervention — The 5-month aerobic exercise intervention is in accordance with the American Heart Association and American College of Sports Medicine physical activity recommendation for optimizing cardiovascular fitness in older adults.Exercise will consist primarily of walking on the treadmill.The goal of the program will be for participants to exercise at a moderate- to high-intensity, defined as 65-80% (ACSM guidelines) of heart rate reserve (HRR), for 30 minutes, 4 days per week.The duration of exercise will progress from 15-20 mins at 50% HRR the 1st week to 30 mins at 65-80% HRR by the end of the 6th week and thereafter.At the start of each session, exercise intensity will be gradually increased to 50% HRR(0.5[HRmax-HRrest]+HRrest)during a 10minute warmup period,and then to the individualized target heart rate training zone for the next 25-30 minutes.Participants will wear a digital heart rate monitoring device for the duration of the training session.

SUMMARY:
This is a small pilot trial of a 5 month aerobic exercise intervention in participants with MCI (n=20) to begin to compare the effects of randomization to use an exercise buddy or to exercise without an assigned buddy. The investigators hypothesize that participants with MCI who exercise with a buddy will have higher adherence to the protocol and greater improvement in 400 meter walk time.

DETAILED DESCRIPTION:
The overall objective of this pilot study is to determine feasibility and gather data that will inform the design of a larger, multicenter, randomized, controlled trial. Specifically, the investigators aim to:

2.1 Determine the feasibility of recruiting persons with MCI and a buddy for an exercise intervention.

- For MCI participants who do not identify a buddy, the investigators will determine the interest and feasibility of recruiting volunteers from the community to be an exercise buddy.

2.2 Determine the effects of having an exercise buddy on:

* adherence to the protocol
* 400 meter walk time, an objective measure of improved physical fitness
* retention and satisfaction for both participant with MCI and buddy

2.3 Establish a scientific partnership with a community based exercise facility.

ELIGIBILITY:
Inclusion Criteria:

Participants:

* Age 60 and up
* Montreal Cognitive Assessment (MoCA) score 16-28
* CDR= 0.5 with memory box at least 0.5.
* Have a person (study partner) who can answer questions about their cognition for the CDR, FAQ and NPI-Q. This should be the same person who will come to all clinic visits whenever possible. This person can be called to answer these questions if unable to come into the clinic.
* Sedentary for past 3 months (< 45 min /wk of exercise, including walking)
* Able to walk 400 meters in < 15 min without assistance
* Willing to exercise 4 days a week at Body Check at CompRehab
* Physician approval for participation in the exercise intervention

Buddy:

* No report of memory problem
* MoCA score > 24 if > HS education; > 23 if 9-12 years; > 22 if ,< 9 years of education

Exclusion Criteria:

Due to Cognitive Confounders:

* Uncontrolled depression (PHQ-9 > 10)
* Schizophrenia or bipolar disorder
* Parkinson's disease
* Hachinski ischemic index > 4
* Daily use of highly anticholinergic medications (such as amitriptyline, diphenhydramine, scopolamine, etc) or benzodiazepines
* Use of stable dose of Cholinesterase inhibitors will be permitted. Must be on a stable dose for 4 weeks.
* Non-English speaking (as we are unable to administer the cognitive tests in languages other than English for this pilot)
* Vitamin B12 deficiency
* Uncontrolled hypothyroidism as measured by TSH blood test

Due to increased risk of or low likelihood of compliance with the exercise program:

* Active ischemic heart disease or angina
* symptomatic heart failure
* stroke
* screening blood pressure SBP > 170 or < 90; DBP > 100 or < 45
* Parkinson's disease or other neurologic disorder that might make exercise on a treadmill or bike unsafe
* Current or planned treatment for cancer
* peripheral artery disease that limits exercise capacity
* Severe respiratory-disease (e.g., COPD) that limits exercise capacity
* Severe arthritis that limits exercise capacity
* Serious conduction disorder, uncontrolled arrhythmia, or new Q waves or ST-segment depressions (> 3 mm) on ECG
* Severe anemia (Hgb < 8)
* Diagnosis of Diabetes and on medication
* Drinks more than 14 alcoholic drinks per week
* Dependent on a cane, walker or other device that would inhibit then from using a treadmill

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adherence (number of sessions attended and exercise duration in targeted heart rate zone) | 4 times a week for 5 months (each exercise session)
  This is a pilot study with the principle outcome measures related to recruitment and retention of participants with MCI and buddies and adherence to the protocol. We are specifically interested in:
  * Time to recruit 20 participants
  * % of participants who identify their own buddy
  * Number of community volunteers to be buddies over the recruitment period
  * Retention at 3- and 5- months
  * Adherence (number of exercise sessions attended, exercise duration in targeted HR zone)

SECONDARY OUTCOMES:
Change in score on Digit Symbol Coding Test | Baseline 3 months and 5 months
Change in 400m walk time (from randomization to 5 months) | Baseline, 3 months and 5 months
Change in Trail Making Test part B score | Baseline and 5 months
change in memory, measured by Rey AVLT delayed recall score, at 5 months | baseline and 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Baker, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States